CLINICAL TRIAL: NCT02919410
Title: Bacterial Colonization With and Without Iodophor-impregnated Adhesive Drapes in Hip Surgery: a Prospective, Randomized Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rothman Institute Orthopaedics (Other)
Responsible Party: Sponsor
Purpose: Prevention
Other Study IDs: JPAR2015
Record Dates: First submitted 2016-09-27; First posted 2016-09-29 (Estimated); Last update posted 2016-09-29 (Estimated); Status verified 2016-09

CONDITIONS: Surgical Wound Infection
MeSH Terms: conditions — Surgical Wound Infection

ARMS (2):
- Surgery performed using iodophor-impregnated adhesive drapes (Active Comparator)
  Interventions: Device: iodophor-impregnated adhesive drapes
- Surgery performed without iodophor-impregnated adhesive drapes (Other)
  Interventions: Other: No adhesive drapes

INTERVENTIONS:
Device: iodophor-impregnated adhesive drapes
  Arms: Surgery performed using iodophor-impregnated adhesive drapes
Other: No adhesive drapes
  Arms: Surgery performed without iodophor-impregnated adhesive drapes

SUMMARY:
This is a prospective, randomized control trial evaluating the efficacy of iodophor-impregnated adhesive drapes for reducing bacterial count in hip surgery.

ELIGIBILITY:
Inclusion Criteria:

* Primary femoroacetabular osteoplasty (FAO) patients
* Primary Periacetabular Osteotomy (PAO) patients

Exclusion Criteria:

* Total hip arthroplasty (THA) patients
* Revision FAO surgery
* Septic or septic arthritis patients
* Patients with systemic or topical allergy to iodine

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2014-10; Primary Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
bacterial count from skin swabs | Immediately post-surgery